CLINICAL TRIAL: NCT07366827
Title: Effectiveness of a Motorized Lumbar Support for Non-specific Low Back Pain: A Randomized Controlled Trial
Brief Title: Effectiveness of Motorised Lumbar Support for Non-specific Low Back Pain
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Corset Saint-Francis (Unknown); MedTeq (Industry)
Responsible Party: Principal Investigator, Hugo Massé-Alarie, Associate Professor, Laval University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2025-3312
Record Dates: First submitted 2026-01-09; First posted 2026-01-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Non-specific Low Back Pain
Keywords: non-specific low back pain; motorized lumbar support; standard lumbar support

STUDY DESIGN:
Who Masked: Participant
Masking Description: The statistician will be blinded to the group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Motorized lumbar support (Experimental): The motorized lumbar support is battery-powered orthosis providing adjustable traction between thoracic and pelvic components, and apply controlled decompressive forces while maintaining mobility.
  Interventions: Other: Motorized lumbar support
- Standard lumbar support (Active Comparator): This is a semi-rigid lumbar support featuring six steel stays, elastic side panels, and a neoprene wrap that allows for individualized adjustment.
  Interventions: Other: Standard lumbar support

INTERVENTIONS:
Other: Motorized lumbar support — Participants will be advised to wear motorized lumbar support for a minimum of 4 hours and a maximum of 8 consecutive hours per day throughout the three-week study period. To reach the target of 4 hours, participants will gradually increase their daily wear time : 2 hours on the first day, 3 hours on the second day and 4 hours on the third day.
  Arms: Motorized lumbar support
Other: Standard lumbar support — Participants will be advised to wear motorized lumbar support for a minimum of 4 hours and a maximum of 8 consecutive hours per day throughout the three-week study period. To reach the target of 4 hours, participants will gradually increase their daily wear time : 2 hours on the first day, 3 hours on the second day and 4 hours on the third day.
  Arms: Standard lumbar support

SUMMARY:
Low back pain (LBP) represents a common musculoskeletal conditions worlwide, causing substantial disability and economic burden. While traditional semi-rigid lumbar supports are commonly prescribed to alleviate LBP symptoms, their effectiveness remains limited by their static mechanical properties and lack of adaptability to movement patterns. Motorized lumbar support offer a novel approach by allowing the application of controlled decompressive forces while maintaining functional mobility. This experimental study aims to compare the effectiveness between a motorized lumbar support and a standard semi-rigid support in adults with non-specific LBP. Seventy adults with non-specific low back pain (LBP) will be recruited. Primary outcomes (pain intensity and physical functioning [daily average]) will be collected daily, while secondary outcomes (average pain intensity over the last week, pain-related disability, etc.) will be assessed at baseline, 3 and 9 weeks after randomization.

DETAILED DESCRIPTION:
LBP represents a common musculoskeletal conditions, causing substantial disability and economic burden. Several strategies, such as education, exercise, manual therapy, psychological techniques and lumbar supports have been recommended for LBP mangement. While traditional semi-rigid lumbar supports are commonly prescribed to alleviate LBP symptoms, their effectiveness remains limited by their static mechanical properties and lack of adaptability to movement patterns. A motorized lumbar support, may offer a novel approach through application of controlled decompressive forces while maintaining functional mobility. An innovative battery-powered orthosis that provides adjustable traction between thoracic and pelvic components, potentially addressing underlying mechanical factors contributing to pain, will be tested in participants with chronic LBP.

This single-blind, parallel-group clinical trial aims to compare the effectiveness of a motorized lumbar support with that of a standard semi-rigid lumbar support in adults suffering from non-specific LBP. Eligible participants will be adults aged 18 to 65 years experiencing LBP with an average pain score of at least 3 out of 10 in the past week, pain related-disability ≥10% at ODI, and pain relief must be present during manual traction (measured by a moderate improvement (+3) on a global rating of change scale. Exclusion criteria include specific spinal pathologies (e.g., fractures, spinal stenosis, cancer), presence of neuropathic pain (leg and back, of 4 at the DN4), pregnancy, high BMI (>32), respiratory and circulatory issues, osteoporosis, recent rib or pelvic fractures, and any contraindications to wearing lumbar supports. A total of 70 participants will be randomly assigned to wear either a motorized lumbar support or a semi-rigid lumbar support . The motorized lumbar support is a battery-powered lumbar orthosis with thoracic and abdominal belts connected by lateral supports. It applies adjustable decompression force to the spine while allowing movement. Each participant will be instructed to wear the assigned support for at least four hours per day over three weeks, excluding while sleeping.

To minimize bias in data collection, subjective variables will be evaluated using REDCap while objective variables will be collectedat research centre. The primary outcomes include daily pain intensity and physical functioning. Secondary subjective outcomes include pain-related disability, average pain intensity of the past week, pain catastrophizing, fear of movement, self-efficacy, acceptability and adverse effects.

The statistician performing the statistical analyses will be blinded to group allocation. Linear mixed models incorporating fixed effects for group (motorized vs. standard support), time, and their interaction, with participants included as a random effect will be used. Daily wearing of the lumbar support, age and self-reported sex will be included as covariates. Intention-to-treat will be used for the main analyses. Per-protocol analyses will be conducted as sensitivity analyses, with the latter including only those who adhered to the recommended usage (minimum 4 hours/day, 5 days/week for 3 weeks). The sample size of 70 participants (35 per group) is planned based on the ability to detect a 2-point difference on the pain scale, with 95% power, a significance level of 0.05, and an estimated 20% dropout rate.

ELIGIBILITY:
Inclusion Criteria

* Adults between 18 and 65 years old with non-specific low back pain.
* Average pain level of ≥3 out of 10 during the previous week.
* Pain-related disability ≥10% at ODI.
* Pain relief must be present during manual traction, measured by a moderate improvement (+3) on a global rating of change scale (anchors: -7 to +7).

Exclusion Criteria:

* Specific cause of low back pain (e.g., fracture, cancer, spinal stenosis, severe spondylolisthesis)
* Presence of neuropathic pain (leg or back of 4 at the DN4).
* Pregnancy.
* Body mass index > 32.
* Waist size between 74 and 115 cm.
* Respiratory and circulatory conditions.
* Osteoporosis.
* Paraplegia and hemiplegia.
* Abdominal wounds at the site of the orthosis.
* Rib or pelvic fractures less than 3 months.
* Presence of electronic medical device.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2027-09-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Pain intensity | Once a day for three weeks.
  The numeric scale from 0 to 10 (0: no pain; 10: worst imaginable pain) will be used to rate average pain intensity experienced during the day.
Physical functioning | Once a day for three weeks.
  The numeric scale from 0 to 10 (0: no difficulty functioning; 10: inability to function) will be used to rate the ability to carry out daily activities.

SECONDARY OUTCOMES:
Pain-related disability | Baseline, week 3 and 9.
  The Oswestry Disability Index (ODI) is a validated and reliable 10-item questionnaire (0 = no disability; 100 = extremely severe disability) recommended for evaluating physical functioning in individuals with LBP.
Pain intensity | Baseline, week 3 and 9.
  The 11-point Numeric Rating Scale (0 = "no pain" to 10 = "the worst pain you can imagine") will be used to measure the average pain intensity over the past week.
Pain catastrophizing | Baseline, week 3 and 9.
  Pain catastrophizing will be evaluated using the Pain Catastrophizing Scale. The Pain Catastrophizing Scale (PCS) is a self-administrated questionnaire of 13 questions measuring catastrophizing thoughts contributing to pain on a 5-point likert scale ranging from 0 ("not at all", low level of catastrophizing thoughts) to 5 ("all the time", high level of catastrophizing thoughts).
Fear of movement | Baseline, week 3 and 9.
  The Tampa Scale of Kinesiophobia is a self-administrated questionnaire used to assess fear of movement using 17 questions on a 4-point scale ranging from 1 ("strongly disagree", low level of kinesiophobia) to 4 ("strongly agree", high level of kinesiophobia).
Pain self-efficacy | Baseline, week 3 and 9.
  Pain self-efficacy will be evaluated using the Pain Self-Efficacy Questionnaire. The Pain Self-Efficacy Questionnaire (PSEQ) is a 10-item questionnaire measuring the confidence people with ongoing pain have in performing activities while in pain, on a 10-point scale from 0 ("not at all confident", low self-efficacy) to 10 ("completely confident", high self-efficacy).
Acceptability | Week 3
  Acceptability of wearing the lumbar support will be evaluated using the Theoretical Framework of Acceptability.
Acceptance | 3 weeks
  Acceptance will be measured using the extended version of the Unified Theory of Acceptance and Use of Technology (UTAUT2).
Adverse events | 3 weeks
  All adverse will be documented and reported.

OTHER OUTCOMES:
Perceived effect of the lumbar support | Once a day for three weeks.
  A "global rating of changes" question type ( "today, what was the effect of wearing the lumbar support") on a 15-point scale (-7 to +7, with -7 = "very great deal worse"; 0 = "no effect" ; +7 = "very great deal better") will be used.
  The perceived effect of the lumbar support will be used only in the per protocol sensitivity analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Hugo Massé-Alarie, PhD, Principal Investigator — Laval University

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (IPD) underlying the results reported in the published article will be made available. The study protocol will also be published.
Supporting Information: Study Protocol
Time Frame: Data will become accessible after the publication and will remain accessible for a period of 5 years after initial release.
Access Criteria: Access to IPD will be granted to qualified researchers whose proposals are methodologically sound and ethically approved. Researchers must obtain approval from their Institutional Review Board (IRB), Research Ethics Board (REB), or equivalent ethics committee, and must sign a Data Use Agreement (DUA) before receiving any data.
  Requests for access should be submitted to: hugo.masse-alarie@fmed.ulaval.ca.